CLINICAL TRIAL: NCT00726232
Title: A Phase 2, Open Label, Dose Regimen Ranging Clinical Study to Determine the Safety and Efficacy of INCB018424 in Patients With Advanced Polycythemia Vera or Essential Thrombocythemia Refractory to Hydroxyurea
Brief Title: Study to Determine the Safety and Efficacy of INCB018424 in Patients With Polycythemia Vera or Essential Thrombocythemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Termination of the clinical trial by sponsor.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-256; Ruxolitinib (Other: Incyte Corporation); 2008-001382-28 (EudraCT Number)
Expanded Access: NCT03147742 (Approved for marketing)
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Myeloproliferative Neoplasm (MPN)
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ruxolitinib 10 mg BID (Experimental): Participants received 10 mg Ruxolitinib orally twice a day (BID) for 56 days (two 28-day cycles) during the dose-ranging phase. After patients completed 2 cycles of treatment at the randomized dose, Investigators were permitted to adjust the dose/regimen on an individual basis to achieve an optimal balance of efficacy and safety. Treatment continued until a patient met a withdrawal criterion, had intolerable toxicity, progression of disease, or withdrew consent.
  Interventions: Drug: Ruxolitinib
- Ruxolitinib 25 mg BID (Experimental): Participants received 25 mg Ruxolitinib orally twice a day (BID) for 56 days (two 28-day cycles) during the dose-ranging phase. After patients completed 2 cycles of treatment at the randomized dose, Investigators were permitted to adjust the dose/regimen on an individual basis to achieve an optimal balance of efficacy and safety. Treatment continued until a patient met a withdrawal criterion, had intolerable toxicity, progression of disease, or withdrew consent.
  Interventions: Drug: Ruxolitinib
- Ruxolitinib 50 mg QD (Experimental): Participants received 50 mg Ruxolitinib orally once a day (QD) for 56 days (two 28-day cycles) during the dose-ranging phase. After patients completed 2 cycles of treatment at the randomized dose, Investigators were permitted to adjust the dose/regimen on an individual basis to achieve an optimal balance of efficacy and safety. Treatment continued until a patient met a withdrawal criterion, had intolerable toxicity, progression of disease, or withdrew consent.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib was administered orally and supplied as 5 mg and 25 mg tablets.
  Other Names: INCB018424

SUMMARY:
To evaluate the safety and efficacy profile of different treatment regimens of Ruxolitinib (INCB018424) administered to two groups of patients; those with polycythemia vera (PV) and those with essential thrombocythemia (ET). Patients in each group were refractory to hydroxyurea or for whom hydroxyurea is contraindicated.

DETAILED DESCRIPTION:
The study consisted of a 2-stage design, which included a dose-ranging phase (during which patients received treatment at their randomized dose) and an expansion phase (after adjustment of dose/regimen to achieve an optimal balance of efficacy and safety). During the dose-ranging phase, patients in each disease group (PV or ET) were randomly assigned in a 1:1:1 ratio independent of each other to receive 1 of 3 treatment regimens with Ruxolitinib, 10 mg twice daily (bid), 25 mg bid, or 50 mg once daily (qd). After patients completed 2 cycles of treatment with Ruxolitinib at the randomized dose, Investigators were permitted to adjust the dose/regimen on an individual basis using their discretion in order to achieve an optimal balance of efficacy and safety. During the expansion phase (ie, after optimization of dose), additional patients with PV or ET were enrolled to receive Ruxolitinib at the dose that was selected upon review of data from the dose-ranging phase. Treatment continued until a patient met a withdrawal criterion, had intolerable toxicity, progression of disease, or withdrew consent.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of polycythemia vera or essential thrombocythemia as determined by treating physician
* Disease refractory to hydroxyurea or for whom treatment with hydroxyurea is contraindicated or have refused further treatment with hydroxyurea due to side effects.
* Patient meets baseline clinical lab parameters

Exclusion Criteria:

* Treatment with interferon alpha or anagrelide within 7 days and hydroxyurea within 1 day of starting INCB018424.
* Patients diagnosed with another malignancy unless the malignancy was cervical intraepithelial neoplasia or basal or squamous cell skin cancer and the patient has been disease free for > 3 years
* Patients receiving therapy with intermediate or high dose steroids greater than the equivalent of 10 mg prednisone per day
* Clinically significant cardiac disease (New York Heart Association (NYHA) Class III or IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-08-20 (Actual); Primary Completion 2010-06-20 (Actual); Study Completion 2018-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Assad, MD, Study Director — Incyte Corporation
Locations (4):
- Houston, Texas, United States
- Italy (3):
  - Bergamo
  - Florence
  - Pavia

REFERENCES:
- [Derived] Pieri L, Pancrazzi A, Pacilli A, Rabuzzi C, Rotunno G, Fanelli T, Guglielmelli P, Fjerza R, Paoli C, Verstovsek S, Vannucchi AM. JAK2V617F complete molecular remission in polycythemia vera/essential thrombocythemia patients treated with ruxolitinib. Blood. 2015 May 21;125(21):3352-3. doi: 10.1182/blood-2015-01-624536. No abstract available. PMID 25999444

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study with 2 sites in the United States and 4 sites in Italy.
Groups:
- Polycythemia Vera (PV): Ruxolitinib 10 mg BID: Participants with Polycythemia Vera received 10 mg Ruxolitinib orally twice a day (BID) for 56 days (two 28-day cycles) during the dose-ranging phase. After patients completed 2 cycles of treatment at the randomized dose, Investigators were permitted to adjust the dose/regimen on an individual basis to achieve an optimal balance of efficacy and safety. Treatment continued until a patient met a withdrawal criterion, had intolerable toxicity, progression of disease, or withdrew consent.
- PV: Ruxolitinib 25 mg BID: Participants with Polycythemia Vera received 25 mg Ruxolitinib orally twice a day (BID) for 56 days (two 28-day cycles) during the dose-ranging phase. After patients completed 2 cycles of treatment at the randomized dose, Investigators were permitted to adjust the dose/regimen on an individual basis to achieve an optimal balance of efficacy and safety. Treatment continued until a patient met a withdrawal criterion, had intolerable toxicity, progression of disease, or withdrew consent.
- PV: Ruxolitinib 50 mg QD: Participants with Polycythemia Vera received 50 mg Ruxolitinib orally once a day (QD) for 56 days (two 28-day cycles) during the dose-ranging phase. After patients completed 2 cycles of treatment at the randomized dose, Investigators were permitted to adjust the dose/regimen on an individual basis to achieve an optimal balance of efficacy and safety. Treatment continued until a patient met a withdrawal criterion, had intolerable toxicity, progression of disease, or withdrew consent.
- Essential Thrombocythemia (ET): Ruxolitinib 10 mg BID: Participants with Essential Thrombocythemia received 10 mg Ruxolitinib orally twice a day (BID) for 56 days (two 28-day cycles) during the dose-ranging phase. After patients completed 2 cycles of treatment at the randomized dose, Investigators were permitted to adjust the dose/regimen on an individual basis to achieve an optimal balance of efficacy and safety. Treatment continued until a patient met a withdrawal criterion, had intolerable toxicity, progression of disease, or withdrew consent.
- ET: Ruxolitinib 25 mg BID: Participants with Essential Thrombocythemia received 25 mg Ruxolitinib orally twice a day (BID) for 56 days (two 28-day cycles) during the dose-ranging phase. After patients completed 2 cycles of treatment at the randomized dose, Investigators were permitted to adjust the dose/regimen on an individual basis to achieve an optimal balance of efficacy and safety. Treatment continued until a patient met a withdrawal criterion, had intolerable toxicity, progression of disease, or withdrew consent.
- ET: Ruxolitinib 50 mg QD: Participants with Essential Thrombocythemia received 50 mg Ruxolitinib orally once a day (QD) for 56 days (two 28-day cycles) during the dose-ranging phase. After patients completed 2 cycles of treatment at the randomized dose, Investigators were permitted to adjust the dose/regimen on an individual basis to achieve an optimal balance of efficacy and safety. Treatment continued until a patient met a withdrawal criterion, had intolerable toxicity, progression of disease, or withdrew consent.
- PV: Ruxolitinib All Doses Combined- Expansion Phase: After the completion of the dose-finding phase of the study, the starting dose of ruxolitinib for the expansion phase was determined to be 10 mg BID for subjects with PV. After subjects completed 8 weeks of ruxolitinib treatment at the starting dose, investigators were permitted to adjust the dose regimen to a maximum total daily dose of 75 mg on an individual basis, using their discretion, in order to achieve an optimal balance of efficacy and safety.
- ET: Ruxolitinib All Doses Combined-expansion Phase: After the completion of the dose-finding phase of the study, the starting dose of ruxolitinib for the expansion phase was determined to be 25 mg BID for subjects with ET. After subjects completed 8 weeks of ruxolitinib treatment at the starting dose, investigators were permitted to adjust the dose regimen to a maximum total daily dose of 75 mg on an individual basis, using their discretion, in order to achieve an optimal balance of efficacy and safety.
Period: Initial Phase (Dose-finding)
Arm/Group | Polycythemia Vera (PV): Ruxolitinib 10 mg BID | PV: Ruxolitinib 25 mg BID | PV: Ruxolitinib 50 mg QD | Essential Thrombocythemia (ET): Ruxolitinib 10 mg BID | ET: Ruxolitinib 25 mg BID | ET: Ruxolitinib 50 mg QD | PV: Ruxolitinib All Doses Combined- Expansion Phase | ET: Ruxolitinib All Doses Combined-expansion Phase
Started | 19 (The starting dose selected for the PV expansion cohort was 10 mg bid hence the sample size is larger) | 8 | 7 | 8 | 22 (The starting dose selected for the ET expansion cohort was 25 mg bid hence the sample size is larger) | 9 | 0 | 0
Safety Evaluable Participants | 19 | 8 | 7 | 8 | 22 | 9 | 0 | 0
ITT Participants | 19 | 8 | 7 | 8 | 22 | 9 | 0 | 0
Completed (Represents participants ongoing treatment.) | 6 | 2 | 2 | 0 | 1 | 0 | 0 | 0
Not Completed | 13 | 6 | 5 | 8 | 21 | 9 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 2 | 1 | 7 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Not completed — Disease progression | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Termination of the trial by sponsor | 4 | 3 | 3 | 4 | 9 | 3 | 0 | 0
Not completed — Per Investigator: lack of response | 1 | 0 | 0 | 2 | 4 | 1 | 0 | 0
Not completed — Unspecified reason | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Expansion Phase
Arm/Group | Polycythemia Vera (PV): Ruxolitinib 10 mg BID | PV: Ruxolitinib 25 mg BID | PV: Ruxolitinib 50 mg QD | Essential Thrombocythemia (ET): Ruxolitinib 10 mg BID | ET: Ruxolitinib 25 mg BID | ET: Ruxolitinib 50 mg QD | PV: Ruxolitinib All Doses Combined- Expansion Phase | ET: Ruxolitinib All Doses Combined-expansion Phase
Started | 0 | 0 | 0 | 0 | 0 | 0 | 34 | 39
Safety Evaluable Participants | 0 | 0 | 0 | 0 | 0 | 0 | 34 | 39
ITT Participants | 0 | 0 | 0 | 0 | 0 | 0 | 34 | 39
Completed (Participants ongoing: last patient last visit (LPLV) occurred 20AUG2018 following the data cutoff.) | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 38
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Not completed — Disease progression | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Termination of the trial by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 16
Not completed — Per Investigator: lack of response | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7
Not completed — Unspecified reason | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety evaluable PV and ET participants.The safety evaluable population included all enrolled participants who received at lease 1 dose of study drug.
Groups:
- PV: Ruxolitinib 10 mg BID: Participants with Polycythemia Vera received 10 mg Ruxolitinib orally twice a day (BID) for 56 days (two 28-day cycles) during the dose-ranging phase. After patients completed 2 cycles of treatment at the randomized dose, Investigators were permitted to adjust the dose/regimen on an individual basis to achieve an optimal balance of efficacy and safety. Treatment continued until a patient met a withdrawal criterion, had intolerable toxicity, progression of disease, or withdrew consent.
- ET: Ruxolitinib 10 mg BID: Participants with Essential Thrombocythemia received 10 mg Ruxolitinib orally twice a day (BID) for 56 days (two 28-day cycles) during the dose-ranging phase. After patients completed 2 cycles of treatment at the randomized dose, Investigators were permitted to adjust the dose/regimen on an individual basis to achieve an optimal balance of efficacy and safety. Treatment continued until a patient met a withdrawal criterion, had intolerable toxicity, progression of disease, or withdrew consent.
- Total: Total of all reporting groups
Arm/Group | PV: Ruxolitinib 10 mg BID | PV: Ruxolitinib 25 mg BID | PV: Ruxolitinib 50 mg QD | ET: Ruxolitinib 10 mg BID | ET: Ruxolitinib 25 mg BID | ET: Ruxolitinib 50 mg QD | Total
Number analyzed (Participants) | 19 | 8 | 7 | 8 | 22 | 9 | 73
Age, Continuous [Mean (Standard Deviation); unit: years]
  Polycythemia vera group | 56.3 (10.98) | 57.0 (11.26) | 51.0 (20.49) | NA (NA) — Age demographic data for the polycythemia vera group. | NA (NA) — Age demographic data for the polycythemia vera group. | NA (NA) — Age demographic data for the polycythemia vera group. | 55.4 (13.20)
  Essential thrombocythemia group | NA (NA) — Age demographic data for the essential thrombocythemia group. | NA (NA) — Age demographic data for the essential thrombocythemia group. | NA (NA) — Age demographic data for the essential thrombocythemia group. | 49.6 (17.89) | 54.1 (11.55) | 52.8 (13.48) | 52.9 (13.19)
Age, Customized [Number; unit: participants]
  >= 65 | 5 | 3 | 2 | 1 | 3 | 3 | 17
  < 65 | 14 | 5 | 5 | 7 | 19 | 6 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 4 | 3 | 13 | 9 | 42
  Male | 8 | 6 | 3 | 5 | 9 | 0 | 31
Hematocrit [Number; unit: participants]
  Hematocrit ≥ 45% | 10 | 7 | 6 | 1 | 4 | 0 | 28
  Hematocrit < 45% | 9 | 1 | 1 | 7 | 18 | 9 | 45
Platelet count [Number; unit: participants]
  ≥400 x 10^9 per liter | 13 | 4 | 6 | 7 | 22 | 9 | 61
  < 400 x 10^9 per liter | 6 | 4 | 1 | 1 | 0 | 0 | 12
White blood cell count [Number; unit: participants]
  ≥ 10 x 10^9 per liter | 12 | 7 | 6 | 2 | 7 | 2 | 36
  < 10 x 10^9 per liter | 7 | 1 | 1 | 6 | 15 | 7 | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Polycythemia Vera Participants With a Confirmed Clinical Partial Response (PR) or Complete Response (CR)
Description: For a confirmed response all criteria must have been sustained for at least 2 months.
  CR:
  * Hematocrit < 45% in men and < 42% in women
  * No phlebotomy for 1 month
  * No palpable splenomegaly
  * White blood cells < 10 x 10^9/L with normal differential and platelets < 400 x 10^9/L
  * No sustained leucopenia or thrombocytopenia (>2 weeks)
  * No systemic PV symptoms (pruritus, night sweats, bone pain, fever, weight loss)
  PR:
  * Hematocrit < 45% in men and < 42% in women
  * 50% reduction in phlebotomy requirements from 6 months before treatment started
  * 50% reduction in palpable splenomegaly
Time Frame: Assessed after 2 cycles (56 days) of treatment on Day 1 of Cycle 3
Population: Polycythemia Vera intent to treat population, including all patients who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | PV: Ruxolitinib 10 mg BID | PV: Ruxolitinib 25 mg BID | PV: Ruxolitinib 50 mg QD
Number analyzed (Participants) | 19 | 8 | 7
percentage of participants | 58 | 50 | 57

2. Secondary Outcome: Percentage of Polycythemia Vera Participants Who Achieved Individual Components of Clinical Response at 12 Weeks
Description: The individual components of clinical response included:
  * Hematocrit (Hct) < 45% without phlebotomy
  * Absence of palpable splenomegaly
  * 50% reduction in spleen size
  * Platelet count ≤ 400 x 10^9/L
  * White blood cell (WBC) count ≤ 10 x 10^9/L
Time Frame: Baseline and Week 12 (Cycle 4, Day 1)
Population: Polycythemia Vera intent to treat population for whom data was available.
Measure: Number; unit: percentage of participants
Arm/Group | PV: Ruxolitinib 10 mg BID | PV: Ruxolitinib 25 mg BID | PV: Ruxolitinib 50 mg QD
Number analyzed (Participants) | 19 | 8 | 7
percentage of participants
  Hematocrit <45% Without Phlebotomy | 95 | 88 | 86
  Absence of palpable splenomegaly | 68 | 50 | 57
  50% reduction in spleen size | 74 | 63 | 86
  Platelet count ≤ 400 x 10^9/L | 58 | 50 | 57
  WBC count ≤ 10 x 10^9/L | 68 | 63 | 43

3. Primary Outcome: Percentage of Essential Thrombocythemia (ET) Participants With a Confirmed Clinical Partial Response (PR) or Complete Response (CR)
Description: For a confirmed response all criteria must have been sustained for at least 2 months.
  Complete Clinical Response:
  * Platelet count < 400 x 10^9/L
  * White blood cell count < 10 x 10^9/L with normal differential and Hematocrit ≤ upper limit of normal
  * Absence of sustained (> 2 weeks) anemia or leucopenia based on institutional normal ranges
  * Absence of systemic ET symptoms (pruritus, bone pain, weakness, night sweats, paresthesias)
  * Absence of palpable splenomegaly
  Partial Clinical Response:
  * Platelet count < 400 x 10^9/L
  * 50% reduction in palpable splenomegaly
Time Frame: Assessed after 2 cycles (56 days) of treatment on Day 1 of Cycle 3.
Population: Essential thrombocythemia intent to treat population, including all patients who took at least 1 dose of study drug. One patient in the 50 mg QD group did not have a response assessment at Cycle 3, Day 1.
Measure: Number; unit: percentage of participants
Arm/Group | ET: Ruxolitinib 10 mg BID | ET: Ruxolitinib 25 mg BID | ET: Ruxolitinib 50 mg QD
Number analyzed (Participants) | 8 | 22 | 8
percentage of participants | 13 | 0 | 0

4. Secondary Outcome: Percentage of Polycythemia Vera Participants Who Achieved Individual Components of Clinical Response at 24 Weeks
Description: as for outcome 2
Time Frame: Baseline and Week 24 (Cycle 7, Day 1)
Population: Polycythemia Vera intent to treat population for whom data was available. 'N' indicates the number of patients for whom data was available for each component.
Measure: Number; unit: percentage of participants
Arm/Group | PV: Ruxolitinib 10 mg BID | PV: Ruxolitinib 25 mg BID | PV: Ruxolitinib 50 mg QD
Number analyzed (Participants) | 19 | 8 | 7
percentage of participants
  Hematocrit <45% Without Phlebotomy | 100 | 88 | 100
  Absence of palpable splenomegaly: number analyzed (Participants) | 18 | 7 | 7
  Absence of palpable splenomegaly | 61 | 43 | 71
  50% reduction in spleen size: number analyzed (Participants) | 18 | 7 | 7
  50% reduction in spleen size | 78 | 71 | 100
  Platelet count ≤ 400 x 10^9/L | 58 | 88 | 86
  WBC count ≤ 10 x 10^9/L | 74 | 25 | 86

5. Secondary Outcome: Percentage of Polycythemia Vera Participants Who Achieved Individual Components of Clinical Response at 36 Weeks
Description: as for outcome 2
Time Frame: Baseline and Week 36 (Cycle 10, Day 1)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | PV: Ruxolitinib 10 mg BID | PV: Ruxolitinib 25 mg BID | PV: Ruxolitinib 50 mg QD
Number analyzed (Participants) | 18 | 8 | 7
percentage of participants
  Hematocrit <45% Without Phlebotomy | 100 | 88 | 100
  Absence of palpable splenomegaly: number analyzed (Participants) | 17 | 7 | 7
  Absence of palpable splenomegaly | 71 | 57 | 86
  50% reduction in spleen size: number analyzed (Participants) | 17 | 7 | 7
  50% reduction in spleen size | 76 | 71 | 100
  Platelet count ≤ 400 x 10^9/L | 67 | 75 | 86
  WBC count ≤ 10 x 10^9/L | 67 | 25 | 71

6. Secondary Outcome: Percentage of Essential Thrombocythemia Participants Who Achieved Individual Components of Clinical Response at 4 Weeks
Description: The individual components of clinical response included:
  * Platelet count ≤ 400 x 10^9/L
  * White blood cell (WBC) count ≤ 10 x 10^9/L
  * 50% reduction in spleen size
  * Absence of palpable splenomegaly
Time Frame: Baseline and 4 weeks (Cycle 2, Day 1)
Population: Essential thrombocythemia intent to treat population. 'N' indicates the number of patients for whom data was available for each component.
Measure: Number; unit: percentage of participants
Arm/Group | ET: Ruxolitinib 10 mg BID | ET: Ruxolitinib 25 mg BID | ET: Ruxolitinib 50 mg QD
Number analyzed (Participants) | 8 | 22 | 9
percentage of participants
  Platelet count ≤ 400 x 10^9/L | 25 | 41 | 33
  WBC count ≤ 10 x 10^9/L | 100 | 100 | 100
  50% reduction in spleen size: number analyzed (Participants) | 6 | 19 | 8
  50% reduction in spleen size | 83 | 95 | 100
  Absence of palpable splenomegaly: number analyzed (Participants) | 6 | 19 | 8
  Absence of palpable splenomegaly | 67 | 89 | 100

7. Secondary Outcome: Percentage of Essential Thrombocythemia Participants Who Achieved Individual Components of Clinical Response at 24 Weeks
Description: as for outcome 6
Time Frame: Baseline and 24 weeks (Cycle 7, Day 1)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | ET: Ruxolitinib 10 mg BID | ET: Ruxolitinib 25 mg BID | ET: Ruxolitinib 50 mg QD
Number analyzed (Participants) | 8 | 22 | 9
percentage of participants
  Platelet count ≤ 400 x 10^9/L: number analyzed (Participants) | 7 | 21 | 8
  Platelet count ≤ 400 x 10^9/L | 14 | 5 | 0
  WBC count ≤ 10 x 10^9/L: number analyzed (Participants) | 7 | 21 | 8
  WBC count ≤ 10 x 10^9/L | 100 | 86 | 100
  50% reduction in spleen size: number analyzed (Participants) | 6 | 19 | 7
  50% reduction in spleen size | 100 | 100 | 100
  Absence of palpable splenomegaly: number analyzed (Participants) | 6 | 19 | 7
  Absence of palpable splenomegaly | 100 | 95 | 100

8. Secondary Outcome: Percentage of Essential Thrombocythemia Participants Who Achieved Individual Components of Clinical Response at 36 Weeks
Description: as for outcome 6
Time Frame: Baseline and 36 weeks (Cycle 10, Day 1)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | ET: Ruxolitinib 10 mg BID | ET: Ruxolitinib 25 mg BID | ET: Ruxolitinib 50 mg QD
Number analyzed (Participants) | 8 | 22 | 9
percentage of participants
  Platelet count ≤ 400 x 10^9/L: number analyzed (Participants) | 7 | 19 | 7
  Platelet count ≤ 400 x 10^9/L | 14 | 11 | 14
  WBC count ≤ 10 x 10^9/L: number analyzed (Participants) | 7 | 19 | 7
  WBC count ≤ 10 x 10^9/L | 100 | 79 | 86
  50% reduction in spleen size: number analyzed (Participants) | 6 | 16 | 6
  50% reduction in spleen size | 100 | 100 | 100
  Absence of palpable splenomegaly: number analyzed (Participants) | 6 | 16 | 6
  Absence of palpable splenomegaly | 100 | 94 | 100

9. Secondary Outcome: Change From Baseline to Week 4 in Polycythemia Vera Symptoms
Description: Patients were asked to rate their symptoms on a scale of 0 (none) to 10 (worse possible) for the prior week giving the worst level of symptoms experienced during the preceding 7 days. A negative change from baseline score indicates improvement in symptoms.
  For patients with Polycythemia Vera, queried symptoms included fever, itching/pruritus, bone pain and night sweats.
Time Frame: Baseline and Week 4 (Cycle 2, Day 1)
Population: Polycythemia Vera intent to treat population who had symptom scores > 0 at baseline for whom data was available.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | PV: Ruxolitinib 10 mg BID | PV: Ruxolitinib 25 mg BID | PV: Ruxolitinib 50 mg QD
Number analyzed (Participants) | 19 | 8 | 7
scores on a scale
  Itching (pruritus): number analyzed (Participants) | 13 | 8 | 5
  Itching (pruritus) | -4.2 (3.63) | -4.6 (1.85) | -2.8 (4.09)
  Bone pain: number analyzed (Participants) | 12 | 2 | 3
  Bone pain | -2.0 (1.95) | -2.5 (0.71) | -4.3 (2.08)
  Fever: number analyzed (Participants) | 2 | 0 | 2
  Fever | -2.0 (1.41) |  | -2.0 (1.41)
  Night sweats: number analyzed (Participants) | 9 | 6 | 3
  Night sweats | -1.9 (2.52) | -2.8 (3.19) | -3.3 (1.15)

10. Secondary Outcome: Change From Baseline to Week 4 in Essential Thrombocythemia Symptoms
Description: Patients were asked to rate their symptoms on a scale of 0 (none) to 10 (worse possible) for the prior week giving the worst level of symptoms experienced during the preceding 7 days. A negative change from baseline score indicates improvement in symptoms.
  For patients with essential thrombocythemia, queried symptoms included itching/pruritus, bone pain, night sweats, paresthesias (tingling or numbness), and weakness.
Time Frame: Baseline and Week 4 (Cycle 2, Day 1)
Population: Essential Thrombocythemia intent to treat population who had symptom scores > 0 at baseline and for whom data was available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ET: Ruxolitinib 10 mg BID | ET: Ruxolitinib 25 mg BID | ET: Ruxolitinib 50 mg QD
Number analyzed (Participants) | 8 | 22 | 8
score on a scale
  Itching (pruritus): number analyzed (Participants) | 3 | 10 | 0
  Itching (pruritus) | -2.7 (2.89) | -1.2 (2.74) |
  Night Sweats: number analyzed (Participants) | 1 | 8 | 3
  Night Sweats | -5.0 (NA) — Only one patient available for this analysis | -1.3 (2.49) | -4.0 (4.36)
  Weakness: number analyzed (Participants) | 3 | 14 | 3
  Weakness | -1.0 (1.00) | -0.2 (2.46) | -1.7 (2.52)
  Bone pain: number analyzed (Participants) | 2 | 13 | 3
  Bone pain | -3.5 (2.12) | -0.4 (2.26) | -2.3 (4.93)
  Paresthesia: number analyzed (Participants) | 3 | 14 | 6
  Paresthesia | -1.7 (2.08) | -1.6 (1.50) | -2.8 (2.93)

11. Secondary Outcome: Change From Baseline to Week 4 in Health-related Quality of Life
Description: Health-related Quality of Life was assessed using the Global Health Status/Quality of Life Scale of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). This scale ranges from 0 to 100, with higher scores indicating higher quality of life.
Time Frame: Baseline and Week 4 (Cycle 2, Day 1)
Population: Intent to treat population. The intent-to-treat (ITT) population included all subjects who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PV: Ruxolitinib 10 mg BID | PV: Ruxolitinib 25 mg BID | PV: Ruxolitinib 50 mg QD | ET: Ruxolitinib 10 mg BID | ET: Ruxolitinib 25 mg BID | ET: Ruxolitinib 50 mg QD
Number analyzed (Participants) | 19 | 8 | 7 | 8 | 22 | 9
units on a scale | 10.9 (10.80) | 6.3 (14.0) | 14.6 (17.78) | -2.1 (10.5) | 3.0 (27.6) | 11.2 (23.4)

ADVERSE EVENTS:
Time Frame: From start of study up to data cutoff at 20 June 2018; approximately 9 years.
Description: Safety evaluable PV and ET participants.The safety evaluable population included all enrolled participants who received at lease 1 dose of study drug.
Arm/Group | PV: Ruxolitinib 10 mg BID | PV: Ruxolitinib 25 mg BID | PV: Ruxolitinib 50 mg QD | ET: Ruxolitinib 10 mg BID | ET: Ruxolitinib 25 mg BID | ET: Ruxolitinib 50 mg QD | PV: Ruxolitinib All Doses Combined- Expansion Phase | ET: Ruxolitinib All Doses Combined-expansion Phase
Serious Adverse Events (participants affected / at risk) | 2/19 | 2/8 | 1/7 | 1/8 | 1/22 | 3/9 | 17/34 | 17/39
Other Adverse Events (participants affected / at risk) | 19/19 | 8/8 | 7/7 | 8/8 | 22/22 | 8/9 | 34/34 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PV: Ruxolitinib 10 mg BID (N=19) | PV: Ruxolitinib 25 mg BID (N=8) | PV: Ruxolitinib 50 mg QD (N=7) | ET: Ruxolitinib 10 mg BID (N=8) | ET: Ruxolitinib 25 mg BID (N=22) | ET: Ruxolitinib 50 mg QD (N=9) | PV: Ruxolitinib All Doses Combined- Expansion Phase (N=34) | ET: Ruxolitinib All Doses Combined-expansion Phase (N=39)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tongue cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestine ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paget's disease of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PV: Ruxolitinib 10 mg BID (N=19) | PV: Ruxolitinib 25 mg BID (N=8) | PV: Ruxolitinib 50 mg QD (N=7) | ET: Ruxolitinib 10 mg BID (N=8) | ET: Ruxolitinib 25 mg BID (N=22) | ET: Ruxolitinib 50 mg QD (N=9) | PV: Ruxolitinib All Doses Combined- Expansion Phase (N=34) | ET: Ruxolitinib All Doses Combined-expansion Phase (N=39)
Anaemia (Blood and lymphatic system disorders) | 16 | 6 | 3 | 5 | 19 | 6 | 27 | 32
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 4 | 1 | 0 | 0 | 0 | 17 | 0
Leukopenia (Blood and lymphatic system disorders) | 4 | 1 | 0 | 0 | 2 | 0 | 8 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Palpitations (Cardiac disorders) | 2 | 0 | 1 | 0 | 4 | 0 | 4 | 6
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myodesopsia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 1 | 1 | 4 | 3 | 12 | 12
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 1 | 3 | 9 | 7
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 2 | 0 | 6 | 3
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 4 | 1 | 4 | 6
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 6 | 5
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dental discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2 | 2 | 4 | 9
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 5
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 4 | 1 | 1 | 2 | 4 | 1 | 13 | 16
Asthenia (General disorders) | 2 | 2 | 0 | 0 | 1 | 1 | 9 | 7
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 2 | 2 | 5 | 5
Oedema peripheral (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 4 | 5
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0
Herpes zoster (Infections and infestations) | 2 | 1 | 1 | 1 | 1 | 1 | 8 | 8
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2 | 0 | 2 | 0 | 9 | 4
Influenza (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0 | 8 | 4
Cystitis (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 1 | 7 | 6
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 1 | 4 | 4
Oral herpes (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 5 | 0
Pharyngitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 3 | 5
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 2 | 1 | 0 | 9 | 11
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 3
Epstein-Barr virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 2 | 1 | 2 | 2 | 5 | 3 | 7 | 14
Blood creatinine increased (Investigations) | 1 | 1 | 1 | 0 | 0 | 2 | 3 | 3
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 4 | 4
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 6 | 2
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 4 | 11
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 3 | 0 | 6 | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 8 | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 1 | 1 | 1 | 11 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 1 | 1 | 8 | 11
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 5 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 4 | 1 | 6 | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 2 | 1 | 1 | 0 | 3 | 0 | 6 | 5
Headache (Nervous system disorders) | 2 | 0 | 1 | 0 | 6 | 2 | 4 | 10
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perineurial cyst (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 2 | 0 | 1 | 1 | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 4 | 1 | 12 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 1 | 1 | 4 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 1 | 1 | 3 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 5 | 4
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucocutaneous rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 6 | 6
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 5 | 8
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cataract operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Serum ferritin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study; provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.